CLINICAL TRIAL: NCT06643962
Title: A Single-Center Prospective Cohort Study to Evaluate the Efficacy and Safety of Intensifying Treatment with Venetoclax in Patients with Newly Diagnosed Acute Myeloid Leukemia (non-APL) and Exhibiting Lower Early Peripheral Blast Clearance Rate After Standard Intensive Induction Chemotherapy
Brief Title: Venetoclax Combined with Intensive Therapy for Acute Myeloid Leukemia Patients with Lower Early Peripheral Blast Clearance Rate After Standard Induction Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TF-IIT-2024-01
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute
Keywords: acute myeloid leukemia; venetoclax; intensive chemotherapy; early peripheral blast clearance; newly diagnosed
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid; Leukemia, Myeloid, Acute | interventions — venetoclax; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assigned interventions (Experimental): Participants with EPBCR>1.5 log (EPBCRhigh) complete the 3+7 regimen and are managed according to standard clinical practice. Participants with EPBCR≦1.5 log (EPBCRlow) receive intensified treatment with venetoclax orally along with the standard 3+7 regimen on days 5-14. A venetoclax dose ramp-up schedule is required in the first induction therapy.
  Interventions: Drug: Venetoclax; Drug: Idarubincin; Drug: Cytarabine

INTERVENTIONS:
Drug: Venetoclax — Venetoclax in the EPBCRlow cohort will be added to the ongoing 3+7 regimen. In the first induction cycle: venetoclax needs to be ramped up: 100 mg on day 5, 200mg on day 6, and 400mg on days 7-14, orally once daily. In the second induction (if required), venetoclax 400mg will be administered orally once daily on days 5-14 without a dose ramp-up schedule. Venetoclax in the EPBCRlow cohort during consolidation therapy: 400mg on days 1-7, orally once daily, along with the consolidation chemotherapy.
  Other Names: Bcl-2 inhibitors
Drug: Idarubincin — Idarubicin (IDA): 10mg/m^2/d (age <60 years old) or 6mg/m^2/d on days 1-3, intravenously (IV).
  Other Names: IDA
Drug: Cytarabine — During induction therapy: 100mg/m2/d on days 1-7, IV. During consolidation therapy: intermediate-dose cytarabine for age >55 years old: 1.0g/m^2 q12h on days 1-3, high-dose cytarabine for age ≦55 years old: 2g/m2 q12h on days 1-3.
  Other Names: Ara-C

SUMMARY:
This single-center prospective cohort study aims to evaluate the efficacy and safety of Intensifying treatment with Venetoclax along with intensive chemotherapy in patients with newly diagnosed acute myeloid leukemia (AML) except acute promyelocytic leukemia (non-APL) and exhibiting lower early peripheral blast clearance rate (EPBCR) after standard Intensive Induction therapy (3+7 regimen).

DETAILED DESCRIPTION:
This is a single-center, prospective cohort study for the intensifying treatment with venetoclax on the standard 3+7 regimen in newly diagnosed AML (non-APL) participants who have lower EPBCR based on ≦1.5log on day 4 of the 3+7 regimen.

The key eligible criteria are newly diagnosed and treatment-naïve AML (non-APL) according to the WHO 2022 criteria. Participants are between 18 and 70 years old and fit for intensive chemotherapy. A leukemia-associated immunophenotype (LAIP) defined by multiparameter flow cytometry (MFC) according to the 2022 ELN recommendation (2022 ELN) is necessary for enrollment in this trial.

All eligible participants receive the 3+7 regimen. Pretreatment with hydroxyurea is permitted to manage leukocytosis.

LAIP+ cells are enumerated on EDTA-anticoagulated peripheral blood collected before chemotherapy on days 1 and 4 of the first induction cycle (each cycle is 28 days). At least 100 circulating LAIP+ cells per microliter on day 1 are required as inclusion criteria to ensure optimal sensitivity. The EPBCR is calculated on day 4 of the first induction regimen as a ratio converted to a logarithmic scale between the absolute peripheral blood LAIP+ cell count on day 1 (baseline) and day 4. A cut-off of 1.5 log is decisional to assign participants to treatment modalities. Participants with EPBCR>1.5 log (EPBCRhigh) complete the 3+7 regimen and are managed according to standard clinical practice. Participants with EPBCR≦1.5 log (EPBCRlow) receive intensified treatment with venetoclax orally along with the standard 3+7 regimen on days 5-14. A venetoclax dose ramp-up schedule is required in the first induction therapy.

After two cycles of induction therapy, participants who fail to achieve composite complete remission (CR/CRi, CRc) may receive an alternative regimen per their physicians' decision.

After CR/CRi is achieved, participants proceed with consolidation therapy or allo-HSCT based on their 2022 ELN risk categories. Participants with favorable risk should go through four cycles (each cycle is 28 days) of consolidation therapy, those with adverse risk should go through allogeneic hematopoietic stem cell transplantation (allo-HSCT) after two cycles of consolidation therapy, and those with intermediate risk can receive allo-HSCT after two cycles of consolidation therapy if suitable donors are available or continue with four cycles of consolidation therapy. Participants receive four cycles of consolidation regimen of intermediate-dose cytarabine for age >60 years old or high-dose cytarabine for age >60 years old. The consolidation therapy will be combined with venetoclax in the EPBCRlow cohort and not in the EPBCRhigh cohort.

After consolidation, participants will receive maintenance therapy per their physicians' decision and be observed.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML, except for the APL subtype, according to the 2022 World Health Organization classification (WHO 2022 criteria)
* Age ≥18 years and ≤70 years
* Eligible for intensive chemotherapy
* No prior chemotherapy for AML except hydroxyurea for up to 14 days during the diagnostic screening phase for the control of peripheral leukemic blasts in patients with leukocytosis (e.g., white blood cell [WBC] counts>25x10^9/L)
* Eastern Cooperative Oncology Group (ECOG) performance status≤2
* Adequate renal function is defined as:

  * Serum creatinine≤2.0×upper limit of normal (ULN)
  * Creatinine clearance (CrCl)>30 mL/min calculated by the Cockcroft-Gault equation.
* Adequate hepatic and heart function is defined as:

  * Serum total bilirubin≤1.5×ULN unless considered due to Gilbert's disease, or leukemic involvement
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP)≤2.5×ULN, unless considered due to leukemic involvement
  * Myocardial enzyme<2.0×ULN
  * Left ventricular ejection fraction is within the normal range by measure of echocardiogram (ECHO)
* Signed a written informed consent form (ICF)
* Female participants who are of non-reproductive potential (i.e., post-menopausal by history of no menses for ≥1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Female participants of childbearing potential must have a negative serum pregnancy test upon study entry

Exclusion Criteria:

* AML with BCR-ABL1 or myeloid blast crisis of CML
* Participants who have received prior treatment for AML with chemotherapy, hypomethylating agents, or venetoclax
* Participants who are ineligible for intensive induction chemotherapy:

  * ≧71 years old OR
  * ≧18 to 70 years old and fulfill at least one criterion associated with lack of fitness for intensive induction chemotherapy:

    * ECOG PS of 2-3
    * Cardiac history of CHF requiring treatment or Ejection Fraction ≦50% or chronic stable angina
    * Diffusing capacity of the lungs for carbon monoxide (DLCO)≦65% or the forced expiratory volume in one second (FEVI) ≦65%
* Participants with a prior history of MDS, MPN, or MDS/MPN
* Participants with other concurrent malignant tumors on treatment, except for:

  * Malignancy treated with curative intent and with no known active disease present for ≧3 years
  * Adequately treated non-melanoma skin cancer or lentigo maligna without current evidence of disease
  * Adequately treated carcinoma in situ without current evidence of disease
  * Localized prostate cancer with a Gleason score of 6 or less
* Pregnant or lactating women
* Active heart disease is defined as any one of the following:

  * Uncontrolled or symptomatic angina pectoris
  * A myocardial infarction six months before enrolled
  * Arrhythmia needs medication or with severe clinical symptoms
  * Uncontrolled or symptomatic congestive heart failure (New York Hear Association [NYHA] classification> grade 2)
* Participants with an active, uncontrolled, systemic fungal, bacterial, or viral infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment
* Participants with an active viral infection caused by HIV, hepatitis B, or hepatitis C virus that cannot be controlled by treatment
* Participants with evidence of central nervous system leukemia before the study treatment
* Participants with epilepsy which needs drug treatment, dementia, or other abnormal mental states that prevent understanding or following the protocol
* Conditions that restrict the intake or absorption of orally administered drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
CRc rate after one cycle of induction therapy | Up to one month
  The proportion of participants achieving CR/CRi by the initiation of next cycle of therapy (each cycle is 28 days).

SECONDARY OUTCOMES:
CRc rate after two cycle of induction therapy | Up to 2 months
  The cumulative proportion of participants achieving CR/CRi after two cycles of induction therapy and before starting the next cycle of therapy.
CRMRD-Rate | Up to 2 months
  The cumulative proportion of participants achieving CR/CRi without measurable residual disease after two cycles of induction therapy and before starting the next cycle of therapy.
Event-free survival (EFS) | Up to 12 months
  The time from enrollment to treatment failure is defined as failure to achieve CR, CRi, or PR after two cycles of induction therapy, death from any cause, or relapse after achieving CR/CRi, whichever occurs first. If no specified events occur at the date of the last disease assessment, participants will be censored.
Relapse free survival (RFS) | Up to 24 months
  From the date of achieving CR/CRi until the date of documented relapse or death due to any cause or the last follow-up day. If no specified events occur at the date of the last disease assessment, participants will be censored.
Overall survival Overall survival (OS) | Up to 24 months
  The time from enrollment to death due to any cause. If death does not occur at the date of the last disease assessment, participants will be censored.

OTHER OUTCOMES:
Baseline genomics | Up to one month
  Genomics at baseline will be assessed at diagnosis using the Next-generation DNA sequencing.
Baseline transcriptomics | Up to one month
  Transcriptomics at baseline will be assessed at diagnosis using the Next-generation RNA sequencing.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No